CLINICAL TRIAL: NCT01766297
Title: Phase II Protocol of Proton Therapy for Partial Breast Irradiation in Early Stage Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Proton Collaborative Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRE007-12
Record Dates: First submitted 2012-12-28; First posted 2013-01-11 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Breast Neoplasm; Breast Tumor; Cancer of the Breast
Keywords: Breast Cancer; Proton; Radiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Radiotherapy (Experimental): Proton Radiotherapy 4.0 Gy (RBE) x10 fractions to 40 Gy (RBE) Total Dose
  Interventions: Radiation: Proton Radiotherapy

INTERVENTIONS:
Radiation: Proton Radiotherapy

SUMMARY:
The purpose of this research study is to compare the effects (good and bad) on women and their cancer using proton radiation therapy.

This study is being done to see if proton radiation therapy will prove to be beneficial for women with early stage breast cancer. A clinical study is necessary to compare the results (good or bad) of proton radiation therapy.

DETAILED DESCRIPTION:
Current standard of care for early stage breast cancer is mastectomy or breast conserving therapy with whole breast irradiation following lumpectomy. However, studies of breast cancer recurrence have demonstrated the majority of tumors to recur in or adjacent to the original tumor site. The question has thus been raised as to whether radiation to the whole breast is necessary or justified. Limiting radiation to the area of the original tumor may reduce acute and long-term skin and organ toxicities while making radiation therapy more convenient and less expensive. Several clinical trials are underway comparing partial breast irradiation (PBI) to whole breast irradiation. Numerous centers are offering partial breast irradiation outside of clinical trials as well, despite the lack of long-term safety and efficacy data on PBI.

Available PBI methods include brachytherapy, in which catheters or balloons are surgically inserted to deliver radiation therapy to the lumpectomy cavity, and conventional external beam radiation therapy, or EBRT. External beam photon therapy is attractive for its non-invasive nature and ability to deliver a more homogenous dose distribution compared to brachytherapy, however it also delivers a greater radiation dose to surrounding normal breast tissue.Proton therapy has the capacity to provide the same advantages as photon EBRT while minimizing dose to normal surrounding tissue. Clinical data on PBI with protons is minimal, however, leaving many questions unanswered. The impetus behind this protocol is to address these gaps by further investigating the feasibility, safety, and efficacy of proton therapy for partial breast irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Must sign study-specific, IRB approved informed consent form prior to study entry. Note consent by legally authorized representative is not allowed for this trial.
* Must be female.
* Must be > = 50 years of age.
* Must have a life expectancy of at least 5 years based on age and co-morbidities.
* Must have pathology proven invasive ductal carcinoma (lobular is not allowed) and/or ductal carcinoma in situ (DCIS).
* One of the following criteria must be met: (a) Tumors that are microscopically multifocal must be 3.0 cm or less in total aggregate size and encompassed within a single scar (b) Patient does not have microscopically multifocal tumor.
* For tumors that are invasive, if in the presence of extensive intraductal component (EIC), the entire pathologic tumor size (including both the intraductal and invasive component) must be 3.0 cm or less.
* Must be Stage 0, I, II (Tis, T1, or T2, N0, M0 per AJCC criteria 7th and/or 8th Ed.). If stage II, the tumor size must be < = 3.0 cm. A patient with invasive histology must have nodal stage pN0 by H&E stains on sentinel node biopsy or axillary lymph node dissection.
* Must have ER positive disease with ER/PR report available.
* For tumors that are invasive, HER2 must be performed (positive or negative is acceptable).
* Must have a lumpectomy performed, with documented negative surgical margins by 0.2 cm or more. If re-excision results in negative surgical margins 0.2 cm or more, patient is eligible.
* If image guidance with daily cone beam CT with direct physician visual assessment is used for treatment positioning, the presence of markers or clips in the surgical bed is recommended but not required. If cone beam CT imaging will NOT be used for image guidance, then the patient must be prepared to have 2 fiducial markers minimum, 3 preferred, placed prior to treatment (if not previously done).

  * If markers or clips were placed at the time of surgery, patient must be able to start treatment within 12 weeks after lumpectomy or re-excision for adequate margins.
  * If markers were not placed at the time of surgery and are needed, patient must have markers placed within 6 weeks after surgery.
  * If systemic chemotherapy was given, patient must have had clips or markers placed at the time of surgery (if they are needed) and patient must have simulation scans within 6 weeks of the completion of the chemotherapy.
* Must be able to start treatment within 12 weeks of surgery or 8 weeks of finalization of chemotherapy.

Exclusion Criteria:

* Previous history of ipsilateral invasive breast cancer or DCIS.
* Any clinical or radiographically suspicious nodes, unless biopsy proven benign.
* Non-epithelial malignancies such as sarcoma or lymphoma.
* Suspicious residual microcalcifications on mammography of either breast, unless negative for malignancy on pathology.
* Multicentric or bilateral disease unless biopsy of the clinical abnormalities are performed and result is negative.
* Lymphovascular space invasion (LVSI) on pathology specimen.
* Any previously treated breast carcinoma or synchronous breast carcinoma in ipsilateral breast.
* Prior radiation therapy to the ipsilateral breast or thorax.
* Paget's disease of the nipple.
* Histologic examination showing invasive lobular histology.
* Skin involvement.
* Breasts technically unsatisfactory for radiation treatment upon the discretion of the treating physician.
* Significant infection or other co-existing medical condition that would preclude protocol therapy such as pregnancy, HIV/AIDS or collagen vascular diseases specifically systemic lupus erythematosus, scleroderma, or dermatomyositis.
* Known BRCA 1 or BRCA 2 mutation.
* Pregnant or lactating.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2013-02; Primary Completion 2027-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
To assess events of freedom from ipsilateral breast recurrence occurrences in patients receiving partial breast proton radiation therapy limited to the region of the tumor. | At 3 years
  Freedom from failure (FFF): The events for FFF will be the first ipsilateral breast cancer recurrence. It is expected that less than 3% of patients will experience an ipsilateral breast cancer recurrence (FFF ≥ 97%). A recurrence rate of ≥ 10% (FFF ≤ 90%) is considered unacceptable. Therefore, the null hypothesis is the FFF of ipsilateral breast cancer recurrence is 90% or lower and the alternative hypothesis is that FFF of ipsilateral breast cancer is 97% or higher.

SECONDARY OUTCOMES:
Assess number and severity of acute and long-term toxicity of partial breast irradiation using proton therapy for the treatment of early stage breast cancer. | On average every 6 months for life
To assess relationship between breast size and partial breast dosimetry. | Average every 6 months for 3 years
Determine quality of life results. | Average every 6 months for 3 years
To determine overall survival rate of patients with breast cancer treated with proton radiation. | At 3 years
To determine recurrence pattern of patients with breast cancer treated with proton partial breast irradiation. | At 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Chang, MD, Study Chair — Proton Collaborative Group
Locations (9):
- United States (9):
  - Mayo Clinic, Scottsdale, Arizona
  - California Protons Cancer Therapy Center, San Diego, California
  - Northwestern Medicine Chicago Proton Center, Warrenville, Illinois
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - McLaren Proton Therapy Center, Flint, Michigan
  - New York Proton Center, New York, New York
  - Oklahoma Proton Center, Oklahoma City, Oklahoma
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Hampton University Proton Therapy Institute, Hampton, Virginia